CLINICAL TRIAL: NCT06230393
Title: An Extension Trial to Evaluate the Long Term Safety and Effectiveness of the STREAMLINE® SURGICAL SYSTEM in Patients With Open-Angle Glaucoma Who Participated in the DF6-CL-20-01 Protocol.
Brief Title: An Extension Trial for Patients With Open-Angle Glaucoma Who Participated in the DF6-CL-20-01 Protocol.
Status: Enrolling by invitation | Type: Observational
Sponsor: New World Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DF6-CL-24-02
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Open Angle Glaucoma; Intraocular Pressure
Keywords: Intraocular Pressure; Glaucoma; MIGS
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: STREAMLINE® SURGICAL SYSTEM — STREAMLINE® SURGICAL SYSTEM

SUMMARY:
The purpose of this study is to evaluate long term safety and effectiveness of the STREAMLINE® SURGICAL SYSTEM

DETAILED DESCRIPTION:
A Retrospective, nonrandomized, open-label study to evaluate the long term safety and IOP-lowering effectiveness of STREAMLINE® SURGICAL SYSTEM in patients with open-angle glaucoma who participated in the DF6-CL-20-01 protocol.

ELIGIBILITY:
Inclusion Criteria:

participated in the DF6-CL-20-01 trial.

Exclusion Criteria:

lost to follow up in the DF6-CL-20-01 trial

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who participated in the DF6-CL-20-01 trial
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in IOP | 24months; 36 months; 48months, 60 months
  From Screening to annual endpoints

SECONDARY OUTCOMES:
Number of IOP lowering medications | 24months; 36 months; 48months, 60 months
  Compared to screening in DF6-CL-20-01 trial

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica 20/20, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No